CLINICAL TRIAL: NCT06536179
Title: New Preclinical and Clinical Approaches to Mesothelioma, an Archetypal Inflammatory Tumor
Brief Title: New Preclinical and Clinical Approaches to Mesothelioma
Status: Recruiting | Type: Observational
Sponsor: Marco Emilio Bianchi (Other)
Collaborators: Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Sponsor-Investigator, Marco Emilio Bianchi, Professor, IRCCS Ospedale San Raffaele
Organization: IRCCS Ospedale San Raffaele (Other)
Other Study IDs: PNRR-TR1-2023-12377199
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study protocol involves the coordination between UO1 (IRCCS San Raffaele Hospital) and UO2 (Istituto Nazionale Tumori di Napoli - IRCCS G. Pascale) to explore the role of HMGB1 and CXCR4 in cancer treatment and metastasis. UO1 focuses on the role of HMGB1 in inflammation, mesothelioma progression, and tissue repair, as well as developing, in future, possible HMGB1 inhibitors for cancer therapy. UO2 specializes in CXCR4's role in cancer, developing CXCR4 antagonists, and tracking CXCR4-dependent metastasis. The hypothesis is that targeting HMGB1 and CXCR4 pathways will inhibit tumor progression and metastasis, enhancing anti-tumor immunity and improving therapeutic outcomes in cancer.

DETAILED DESCRIPTION:
This is a multicentric cross-sectional observational study with an additional blood volume collected during blood sampling performed for normal clinical practice. The enrollment will take

ELIGIBILITY:
Inclusion Criteria:

* Patients with Mesothelioma:

Clinical suspicion or histologically confirmed diagnosis of pleural mesothelioma.

* Candidates for surgical intervention.
* Age 18 years or older. It is possible to include both male and female patients, male and female patients of reproductive age, as well as breastfeeding women.
* Capacity to comprehend the study nature and provide autonomously informed consent.

Control Group patients:

* Absence of pleural mesothelioma but presence of other histologically confirmed diseases (neoplastic, inflammatory, or infectious).
* Candidates for surgical intervention.
* Age 18 years or older. It is possible to include both male and female patients, male and female patients of reproductive age, as well breastfeeding women.
* Ability to understand the study nature and provide autonomously informed consent.

If the patient's diagnosis, whether provisional or definitive, does not confirm the clinical suspicion, they will not undergo further evaluation in the study.

Exclusion Criteria:

* Lack of biopsy material.
* pregnancy.
* Unwillingness to sign the Informed Consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For this study, San Raffaele Hospital and Istituto Nazionale Tumori IRCCS Fondazione G. Pascale will enroll both:
  * patients with a clinical suspicion of mesothelioma (cancer patients), and for which surgery is indicated and will be performed as per clinical practice. From the biopsies thus obtained in accordance with normal clinical practice (the biopsies provided to us by the clinic are considered waste material) whose biopsies mesothelioma organoids will be obtained;
  * patients with a clinical suspicion or diagnosis different from that of mesothelioma, from whose biopsies (the biopsies provided to us by the clinic are considered waste material) non-tumoral organoids will be obtained to serve as controls for the tumoral ones.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
To set up spheroids models to study and serve as a platform | 0/baseline
  Number of spheroids with infiltrated macrophages. About of 30% of macrophages infiltrated into spheroids.
To set up spheroids models and serve as a platform | 0/baseline
  Evaluation of macrophages polarization status M1 or M2 based on different genes and proteins expression using qPCR and Flow Cytometry.
To set up organoid models | 0/baseline
  Number of organoids formation. About of 30% of biopsies generated organoids.
Test inhibitors on spheroids and organoids and assess the response of individual patients to therapy | 0/baseline
  Rate of growth to test the efficacy of anti-CSF1R, BoxA and DFL using human mesospheres from MPM primary cell lines derived from patients and monocytes from controls.

SECONDARY OUTCOMES:
To investigate inhibitors of the CXCR4-CXCL12-HMGB1 axis on the crosstalk | 0/baseline
  Percentage of migrated or invaded MPM cell lines NCI-H2052 (BAP1 WT/NF2 MUT) vs NCI-H28 (BAP1 mut/NF2 WT) with and without macrophages in presence of CDDP-Nivolumab (NIVO)-Peptide R54.
To investigate inhibitors of the CXCR4-CXCL12-HMGB1 axis on the crosstalk | 0/baseline
  Percentage of cell death of Tregs/Macrophages from peripheral blood and pleural effusion derived from MPM patients treated with and without R54.
To investigate inhibitors of the CXCR4-CXCL12-HMGB1 axis on the crosstalk | In vivo experiment 3 weeks.
  Overall survival of mice with MPM treated with CDDP-anti-PD-1/R54.

OTHER OUTCOMES:
Repurposing Diflunisal as antitumor drug in MPM | In vivo experiment 3 weeks.
  Overall survival of MPM mice treated with DFL in combination with the gold-standard treatment of MM patients, i.e. checkpoint inhibitors (Nivolumab + Ipilimumab).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bianchi, Professor, Principal Investigator — IRCCS Ospedale San Raffaele; Vincenzo Sforza, MD, Principal Investigator — Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale
Locations (2):
- Italy (2):
  - Istituto Nazionale Tumori IRCCS Fondazione G.Pascale, Napoli, Campania
  - IRCCS San Raffaele, Milan, Lombardy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shimizu Y, Dobashi K, Imai H, Sunaga N, Ono A, Sano T, Hikino T, Shimizu K, Tanaka S, Ishizuka T, Utsugi M, Mori M. CXCR4+FOXP3+CD25+ lymphocytes accumulate in CXCL12-expressing malignant pleural mesothelioma. Int J Immunopathol Pharmacol. 2009 Jan-Mar;22(1):43-51. doi: 10.1177/039463200902200106. PMID 19309551
- [Background] Bianchi ME, Crippa MP, Manfredi AA, Mezzapelle R, Rovere Querini P, Venereau E. High-mobility group box 1 protein orchestrates responses to tissue damage via inflammation, innate and adaptive immunity, and tissue repair. Immunol Rev. 2017 Nov;280(1):74-82. doi: 10.1111/imr.12601. PMID 29027228
- [Background] Santagata S, Napolitano M, D'Alterio C, Desicato S, Maro SD, Marinelli L, Fragale A, Buoncervello M, Persico F, Gabriele L, Novellino E, Longo N, Pignata S, Perdona S, Scala S. Targeting CXCR4 reverts the suppressive activity of T-regulatory cells in renal cancer. Oncotarget. 2017 Aug 19;8(44):77110-77120. doi: 10.18632/oncotarget.20363. eCollection 2017 Sep 29. PMID 29100374
- [Background] Li B, Zeng Y, Reeves PM, Ran C, Liu Q, Qu X, Liang Y, Liu Z, Yuan J, Leblanc PR, Ye Z, Sluder AE, Gelfand JA, Brauns TA, Chen H, Poznansky MC. AMD3100 Augments the Efficacy of Mesothelin-Targeted, Immune-Activating VIC-008 in Mesothelioma by Modulating Intratumoral Immunosuppression. Cancer Immunol Res. 2018 May;6(5):539-551. doi: 10.1158/2326-6066.CIR-17-0530. Epub 2018 Mar 6. PMID 29511032
- [Background] Kinoshita Y, Hamasaki M, Yoshimura M, Matsumoto S, Iwasaki A, Nabeshima K. Hemizygous loss of NF2 detected by fluorescence in situ hybridization is useful for the diagnosis of malignant pleural mesothelioma. Mod Pathol. 2020 Feb;33(2):235-244. doi: 10.1038/s41379-019-0309-6. Epub 2019 Jun 23. PMID 31231129
- [Background] D'Alterio C, Buoncervello M, Ierano C, Napolitano M, Portella L, Rea G, Barbieri A, Luciano A, Scognamiglio G, Tatangelo F, Anniciello AM, Monaco M, Cavalcanti E, Maiolino P, Romagnoli G, Arra C, Botti G, Gabriele L, Scala S. Targeting CXCR4 potentiates anti-PD-1 efficacy modifying the tumor microenvironment and inhibiting neoplastic PD-1. J Exp Clin Cancer Res. 2019 Oct 28;38(1):432. doi: 10.1186/s13046-019-1420-8. PMID 31661001
- [Background] Zhang M, Luo JL, Sun Q, Harber J, Dawson AG, Nakas A, Busacca S, Sharkey AJ, Waller D, Sheaff MT, Richards C, Wells-Jordan P, Gaba A, Poile C, Baitei EY, Bzura A, Dzialo J, Jama M, Le Quesne J, Bajaj A, Martinson L, Shaw JA, Pritchard C, Kamata T, Kuse N, Brannan L, De Philip Zhang P, Yang H, Griffiths G, Wilson G, Swanton C, Dudbridge F, Hollox EJ, Fennell DA. Clonal architecture in mesothelioma is prognostic and shapes the tumour microenvironment. Nat Commun. 2021 Mar 19;12(1):1751. doi: 10.1038/s41467-021-21798-w. PMID 33741915
- [Background] Bertolini G, Cancila V, Milione M, Lo Russo G, Fortunato O, Zaffaroni N, Tortoreto M, Centonze G, Chiodoni C, Facchinetti F, Pollaci G, Taie G, Giovinazzo F, Moro M, Camisaschi C, De Toma A, D'Alterio C, Pastorino U, Tripodo C, Scala S, Sozzi G, Roz L. A novel CXCR4 antagonist counteracts paradoxical generation of cisplatin-induced pro-metastatic niches in lung cancer. Mol Ther. 2021 Oct 6;29(10):2963-2978. doi: 10.1016/j.ymthe.2021.05.014. Epub 2021 May 21. PMID 34023505
- [Background] Oien DB, Sarkar Bhattacharya S, Chien J, Molina J, Shridhar V. Quinacrine Has Preferential Anticancer Effects on Mesothelioma Cells With Inactivating NF2 Mutations. Front Pharmacol. 2021 Sep 21;12:750352. doi: 10.3389/fphar.2021.750352. eCollection 2021. PMID 34621176
- [Background] Santagata S, Rea G, Castaldo D, Napolitano M, Capiluongo A, D'Alterio C, Trotta AM, Ierano C, Portella L, Di Maro S, Tatangelo F, Albino V, Guarino R, Cutolo C, Izzo F, Scala S. Hepatocellular carcinoma (HCC) tumor microenvironment is more suppressive than colorectal cancer liver metastasis (CRLM) tumor microenvironment. Hepatol Int. 2024 Apr;18(2):568-581. doi: 10.1007/s12072-023-10537-6. Epub 2023 May 4. PMID 37142825
- [Background] Husain AN, Colby T, Ordonez N, Krausz T, Attanoos R, Beasley MB, Borczuk AC, Butnor K, Cagle PT, Chirieac LR, Churg A, Dacic S, Fraire A, Galateau-Salle F, Gibbs A, Gown A, Hammar S, Litzky L, Marchevsky AM, Nicholson AG, Roggli V, Travis WD, Wick M; International Mesothelioma Interest Group. Guidelines for pathologic diagnosis of malignant mesothelioma: 2012 update of the consensus statement from the International Mesothelioma Interest Group. Arch Pathol Lab Med. 2013 May;137(5):647-67. doi: 10.5858/arpa.2012-0214-OA. Epub 2012 Aug 28. PMID 22929121